CLINICAL TRIAL: NCT04910581
Title: Inhibitory rTMS Applied on Laryngeal Motor Cortex in Wilson's Disease Patients With Dysarthria
Brief Title: rTMS in Wilson Disease Dysarthria
Acronym: WILSTIM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D20180404
Record Dates: First submitted 2021-05-14; First posted 2021-06-02 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Wilson Disease
Keywords: dyasarthria, repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Intervention Model Description: After randomization, patients are to receive blindly the first rTMS session according to the arm (placebo or active). A second stimulation session is to be performed 3 days apart to apply the reverse arm.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients are centrally randomized to receive first either the active stimulation (80% of the resting motor threshold) or the sham stimulation (using a visually identical coil to reproduce the click sound and the scalp sensation of the active coil). The operator is unblided. The evaluator is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental stimulation (Active Comparator): Patients receive an inhibitor treatment of rTMS using activ coil (MCF B65 coil) for 30 minutes at 1Hz at 80% of the resting motor threshold (MagPro stimulator; MagVenture A / S, Farum, Denmark) onto the left laryngeal cortex located thanks to a neuronavigation device (Syneika one [SYN1], Syneika, Cesson-Sévigné, France).
  Interventions: Procedure: rTMS
- Sham stimulation (Placebo Comparator): Patients receive a treatment of rTMS using placebo coil (MCF P B65 coil) for 30 minutes at 1Hz (MagPro stimulator; MagVenture A / S, Farum, Denmark) onto the left laryngeal cortex located thanks to a neuronavigation device (Syneika one [SYN1], Syneika, Cesson-Sévigné, France).
  Interventions: Procedure: Sham stimulation

INTERVENTIONS:
Procedure: rTMS — Single 30-minutes session of 1Hz rTMS applied over the left laryngeal motor cortex
  Arms: Experimental stimulation
Procedure: Sham stimulation — Single 30-minutes session of sham stimulation applied over the left laryngeal motor cortex
  Arms: Sham stimulation

SUMMARY:
Wilson disease is a hereditary hepatic and neurological disease associated with copper accumulation. Neurological symptoms are of extra-pyramidal, cerebellar and dystonic origin. Dysarthria is one of the debilitating symptoms of Wilson disease poorly responsive to pharmacological treatment. The most common form is a dystonic hyperkinetic Dysarthria.

Pathophysiology of dystonia is still not elucidated. Motor cortex hyperexcitability has been demonstrated in various forms of dystonia. Furthermore, rTMS inhibitory applied over motor cortex has been shown to transitory reduce dystonic symptoms in various forms of dystonia.

In the present study, we investigate the effect of a single 1Hz 20-minutes inhibitory rTMS session applied over the motor laryngeal cortex on dyasarthria is the main kinetic dysarthria has been shown to be associated with inhibition of laryngeal motor cortex in Parkinson disease.

DETAILED DESCRIPTION:
A consecutive series of Wilson disease patients with dystonic hyperkinetic dysarthria will be prospectively recruited.

Patients will receive 3 days apart to two rTMS sessions.

rTMS procedures will be performed with a figure of eight coiled. A single 20-minutes 1 Hz biphasic stimulation (1200 pulses) session will be applied over the laryngeal motor cortex. A brain imaging positioning device will be used during all the procedure A second stimulation session will be performed 3 days apart.

Patients will be centrally randomized to receive first either the active stimulation (80% of the resting motor threshold) or the sham stimulation (using a visually identical coil to reproduce the click sound and the scalp sensation of the active coil).

A TMS evaluation of cortical silent period over the left motor cortex will be performed before the first rTMS session.

Before and immediately after each stimulation (active or sham) patient will received an clinical evaluation including Clinical Assessment Battery for Dysarthria intelligibility score, "A" phonation time, diadococinesia , bucco-linguo-facial motricity score and UWDRS.

A standard 20-minutes EEG will be performed before the first rTMS session and immediately after the second rTMS session.

ELIGIBILITY:
Inclusion Criteria:

* Conseting adult patients with social insurance
* Wilson disease with dystonic hyperkinetic dysarthria
* Stable pharmacological therapy n the last 6 monts
* Brain MRI in the previous 6 months, without additional brain lesion
* Patients that did not receive botulinium toxin in the previous 4 months

Exclusion Criteria:

* Incapacitated adult
* Previous mdedical history of epilepsia
* Pregnancy or breastfeeding
* Brain lesion outside basal ganglia on brain MRI
* Patient consider by the investigator not able to sustain an 30 minutes rTMS session without moving
* Vocal chord lesion
* Previous history of laryngeal surgery
* rTMS contra indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Improvement of the Clinical Assessment Battery for Dysarthria intelligibility score | within 30 minutes after stimulation session at Day1 and Day4
  Improvement of the Clinical Assessment Battery for Dysarthria intelligibility score with active stimulation in comparison to sham stimulation

SECONDARY OUTCOMES:
Improvement of the Clinical Assessment Battery for Dysarthria intelligibility sub-scores | within 30 minutes after stimulation session at Day1 and Day4
  Improvement of the Clinical Assessment Battery for Dysarthria intelligibility sub-scores with active stimulation in comparison to sham stimulation
the "A" phonation time | within 30 minutes after stimulation session at Day1 and Day4
  Improvement of the "A" phonation time with active stimulation in comparison to sham stimulation
Improvement of the diadococinesia | within 30 minutes after stimulation session at Day1 and Day4
  Improvement of the diadococinesia with active stimulation in comparison to sham stimulation
Improvement of text reading | within 30 minutes after stimulation session at Day1 and Day4
  Improvement of text reading with active stimulation in comparison to sham stimulation
Improvement of bucco-linguo-facial motricity | within 30 minutes after stimulation session at Day1 and Day4
  Improvement of bucco-linguo-facial motricity with active stimulation in comparison to sham stimulation
Improvement bucco-linguo-facial motricity | within 30 minutes after stimulation session at Day1 and Day4
  Improvement bucco-linguo-facial motricity with active stimulation in comparison to sham stimulation
Correlation between clinical Assessment Battery for Dysarthria intelligibility score and UWDRS, and MRI brain atrophy and basal ganglia lesions | at Day1 and Day4
  Correlation of changes in the Battery for Dysarthria intelligibility score with clinical parameters (age at diagnosis, delay related to first symptoms, degree of neurological handicap and brain lesions observed on basline MRI (cortical atrophy and lesions of the basal ganglia)
Side effects of rTMS | within few hours after stimulation session at Day1 and Day4
  Any side effect after stimulation (fatigue, neck pain, neck stiffness, dizziness, nausea, itching, mood disorders ..) will be collected following the stimulation.
  Side effects of rTMS are rare. Most often they are minor and transient.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service de Physiologie Clinique-Explorations Fonctionnelles, AP-HP, Hôpital Lariboisière, Paris
  - Service de Neurologie, Hopital Fondation Adolphe de Rothschild, Paris

IPD SHARING:
Plan to Share IPD: No